CLINICAL TRIAL: NCT00006028
Title: Evaluation of Gemcitabine and Cisplatin in Recurrent, Platinum Resistant and Refractory Ovarian Cancer
Brief Title: Gemcitabine Plus Cisplatin in Treating Patients With Ovarian Epithelial Cancer or Primary Peritoneal Cancer That Is Recurrent or Has Not Responded to Platinum-based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000068041; GOG-0126L
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2003-03

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine plus cisplatin in treating patients who have primary ovarian epithelial cancer or primary peritoneal cancer that is recurrent or has not responded to platinum-based chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the anti-tumor activity of gemcitabine and cisplatin in patients with recurrent or refractory platinum-resistant ovarian epithelial cancer or primary peritoneal carcinoma who have failed on higher priority treatment protocols.
* Determine the nature and degree of toxicity of this regimen in this patient population.
* Correlate ex vivo drug sensitivity and resistance with clinical response to this regimen in these patients.
* Correlate molecular markers of drug responsiveness and cellular apoptosis with ex vivo measures of drug resistance in these patients.

OUTLINE: This is a multicenter study.

Patients receive cisplatin IV over 1 hour followed by gemcitabine IV over 1 hour on days 1 and 8. Courses repeat every 4 weeks in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 5-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary ovarian epithelial cancer or primary peritoneal carcinoma

  * Recurrent or persistent disease
* Bidimensionally measurable disease by physical examination or medical imaging techniques

  * Sonography is acceptable if lesions are clearly defined on initial examination and bidimensionally measurable
  * Ascites and pleural effusions are not considered measurable disease
* Must not be eligible for a higher priority Gynecologic Oncology Group protocol
* Must have received one, and only one, prior platinum-based chemotherapy regimen containing carboplatin, cisplatin, or another organoplatinum compound for management of primary disease

  * Initial treatment may include high-dose therapy, consolidation, or extended therapy administered after surgical or nonsurgical assessment
  * If no prior paclitaxel, a second regimen containing paclitaxel allowed
* Platinum-resistant or refractory (i.e., treatment-free interval after platinum-based therapy of less than 6 months or progressed during platinum-based therapy)

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* Sensory and motor neuropathy no greater than grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic or immunologic therapy for ovarian or peritoneal cancer

Chemotherapy:

* See Disease Characteristics
* No other prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimens
* No prior gemcitabine
* At least 3 weeks since prior chemotherapy for ovarian or peritoneal cancer and recovered

Endocrine therapy:

* At least 1 week since prior hormonal therapy for ovarian or peritoneal cancer
* Concurrent continuation of hormonal replacement therapy allowed

Radiotherapy:

* At least 3 weeks since prior radiotherapy for ovarian or peritoneal cancer and recovered
* No prior radiotherapy to only site of measurable disease
* No prior radiotherapy to more than 25% of bone marrow

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior surgery for ovarian or peritoneal cancer and recovered

Other:

* At least 3 weeks since other prior therapy for ovarian or peritoneal cancer
* No prior cancer treatment that would preclude study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-01; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A. Brewer, MD, Study Chair — University of Illinois College of Medicine at Peoria
Locations (31):
- United States (30):
  - Community Hospital of Los Gatos, Los Gatos, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Ellis Fischel Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - CCOP - M.D. Anderson Research Base, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Brewer CA, Blessing JA, Nagourney RA, Morgan M, Hanjani P. Cisplatin plus gemcitabine in platinum-refractory ovarian or primary peritoneal cancer: a phase II study of the Gynecologic Oncology Group. Gynecol Oncol. 2006 Nov;103(2):446-50. doi: 10.1016/j.ygyno.2006.03.018. Epub 2006 Apr 27. PMID 16643994